CLINICAL TRIAL: NCT02760589
Title: Clinical Evaluation After Anterior Cruciate Ligament Tears (Internal Brace Technique vs. ACL Reconstruction vs. Conservative Treatment) With Special Regard to Magnetic Resonance Imaging and Functional Performance
Brief Title: Magnetic Resonance Imaging and Functional Performance Outcome After ACL Repair With Internal Brace Technique
Status: Completed | Type: Observational
Sponsor: AUVA (Other)
Responsible Party: Principal Investigator, Georg Mattiassich, Dr. med. unit., AUVA
Other Study IDs: 7/2015
Record Dates: First submitted 2015-11-27; First posted 2016-05-03 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: ACL tear; ACL lesion; ACL reconstruction; InternalBrace; functional performance test; anterior cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ACL tear - conservative: conservative treatment
- ACL tear - ACL reconstruction: reconstruction of the ACL with autologous tendons
- ACL tear - Internal brace: augmentation of the ruptured ACL with Internal brace
- healthy subjects: control group of healthy subjects with no previous injury

SUMMARY:
The purpose of the study is a clinical evaluation with special regard to magnetic resonance imaging and functional performance at least one year after injury / surgery in all three groups (subjects who underwent InternalBrace surgery, subjects who underwent surgery with a semitendinosus graft and subjects who were treated conservatively).

DETAILED DESCRIPTION:
Lesions of the anterior cruciate ligament (ACL) are the most common ligamentous injuries with an increasing incidence. 77% of ACL insufficient knees result in moderate to high physical limitations. Different surgical treatments have been described. ACL reconstruction with either a semitendinosus or patella tendon graft is regarded as the gold standard of operative therapy. Despite numerous studies representing good and excellent outcome after ACL reconstruction, a recent Meta-analysis of Biau et al. 2006 revealed that only 40% of patients gain full functional recovery.

Since the native ACL is considered to be an important factor for the proprioceptive sensation, a removal during the reconstruction might have an adverse influence on muscular stabilisation, rehabilitation and functional performance of the knee joint. Thus a primary repair of the native ACL seems reasonable.

For tears of the anterior cruciate ligament near the femoral attachment a new method of surgical treatment can be applied. The InternalBrace method by Arthrex is performed arthroscopically and involves reattaching of the ACL that has avulsed off the femoral wall using a FiberTape by Arthrex. To the authors knowledge the augmentation with FiberTape by Arthrex has not been systematically evaluated. Promising results have been presented recently using a comparable method, which showed a high patient satisfaction, faster rehabilitation and a high rate of return to pre-injury sports level.

To assess the functional performance, a further aim of the study is to develop a new test battery consisting of strength tests and single-leg hop tests with the ability to distinguish between the functional performance of the injured and the uninjured leg in patients with ACL deficiency. Test batteries consisting of several hop tests has been described in the previous literature indicating a good test-retest reliability measuring lower leg performance. The functional performance is defined using the limb symmetry index in percent between each individuals lower limbs. This study aims to determine the LSI of healthy subjects using the values achieved by the subjects in the control group. A limb symmetry index (LSI) between 85% and 95% is considered sufficient for return to pivoting sports in patients after knee injury.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects
* Age between 18 and 60 years
* Patients who sustained an isolated rupture of the anterior cruciate ligament at least 12 month after injury (for the subjects who received conservative therapy), respectively surgery (for the two groups in which subjects underwent surgery)
* MRI-confirmed tear of the anterior cruciate ligament near the femoral attachment
* Surgical treatment of the InternalBrace group must have been performed within the first six weeks after injury
* Women of reproductive age
* Confirmed written consent of each subject

Exclusion Criteria:

* Injury to the other knee
* Previous knee injuries which required treatment
* Concomitant injuries such as fractures, articular cartilage lesions reaching subchondral bone, meniscal tears or lesions of the collateral ligaments which required an additional surgical intervention and therefore an extended post-op rehabilitation protocol
* Pregnant and nursing women
* Claustrophobia
* Existing contraindication against performing an MRI scan
* Taking certain concomitant medication(s) (especially cortisone), or conditions that interfere with a patient's ability to comply with all procedures
* Circumstances that interfere with the participant's ability to give informed consent (diminished understanding or comprehension, or a language other than German or English spoken

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with rupture of the ACL between 18 and 60 years
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Signal Intensity in Magnetic resonance Imaging | at least one year after injury
  The integration of the ligament in magnetic resonance imaging is represented by using values from 1 to 3 (1= continuous ligament; 2= wavy but continuous ligament contour; 3= non-delineated ligament) which are determined by an experienced independent radiologist. Source of the data: axial, coronal, and sagittal scans with proton density-weighted sequences with and without fat saturation by a 1.5-Tesla MRI unit (1.5-Tesla MRI unit, Espree; Siemens AG, Erlangen, Germany).

SECONDARY OUTCOMES:
Limb symmetry Index | at least one year after Injury / surgery
  The functional performance is defined using the LSI in percent between each individual's lower limbs using a diagnostic battery. The test battery consists of a standardized warm-up protocol followed by an isometric strength test (testing the maximum voluntary isometric contraction) of the hamstrings in prone position in 90 degree knee flexion using a portable dynamometer (Mecmesin Advanced Force Gauge, Mecmesin, UK), which is attached to a wall bar with a non-stretchable rope. After that several single-leg jump tests are performed: (1) single-leg hop for distance, (2) single-leg 6m timed hop, (3) single-leg triple crossover hop for distance and (4) side hop test. Finally, a fatigued single-leg hop for distance is conducted following a fatigue protocol consisting of alternating squat lunges to exhaustion for the duration of two minutes. The LSI will be calculated for the best trial in each of the five hop tests and for the overall combination as an average of the hop tests.
Subjective Outcome: German Version of the IKDC Subjective Knee Form (International Knee Documentation Committee | at least one year after Injury
  Source of the data: knee evaluation form Results: continuous data between 0 and 100
Subjective Outcome: German Version of the WOMAC (Western Ontario and McMaster Universities Arthritis Index | at least one year after Injury
  Source of the data: 5-point Likert-type of a subjective patient questionnaire of 24 items divided into 3 subscales (pain: 5 items, stiffness: 2 items, physical function: 17 items) Result: ordinal data (pain=0-20, stiffness=0-8, physical function=0-68)
Subjective Outcome: SF-12 (short form) | at least one year after Injury
  Source of the data: 5-point Likert-type of a subjective patient questionnaire of 12 items Result: continuous data between 0 and 100 (the higher the number, the better the subjective physical and mental health)
Subjective Outcome: German Version of the KOOS (Knee Osteoarthritis Outcome Score) | at least one year after Injury
  Source of the data: patient-administered subjective questionnaire of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL) What form the data will take: a normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Subjective Outcome: German Version of the modified Lysholm-Score by Lysholm and Gillquist | at least one year after Injury
  Source of the data: 8-item patient-administered questionnaire Result: continuous data between 0 and 100
Subjective Outcome: German Version of the TAS (Tegner activity scale) | at least one year after Injury
  The physical activity level of all subjects in all groups is estimated with the German Version of the TAS (Tegner activity scale).
  Source of the data: patient questionnaire Result: ordinal data between 0 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Georg Mattiassich, MD, Principal Investigator — AUVA
Locations (1):
- Traumacenter Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Individual data may be allocated confidentially to each individual at the end of the investigation.

REFERENCES:
- [Background] Siegel L, Vandenakker-Albanese C, Siegel D. Anterior cruciate ligament injuries: anatomy, physiology, biomechanics, and management. Clin J Sport Med. 2012 Jul;22(4):349-55. doi: 10.1097/JSM.0b013e3182580cd0. PMID 22695402
- [Background] Engebretsen L, Benum P, Fasting O, Molster A, Strand T. A prospective, randomized study of three surgical techniques for treatment of acute ruptures of the anterior cruciate ligament. Am J Sports Med. 1990 Nov-Dec;18(6):585-90. doi: 10.1177/036354659001800605. PMID 2285086
- [Background] Biau DJ, Tournoux C, Katsahian S, Schranz PJ, Nizard RS. Bone-patellar tendon-bone autografts versus hamstring autografts for reconstruction of anterior cruciate ligament: meta-analysis. BMJ. 2006 Apr 29;332(7548):995-1001. doi: 10.1136/bmj.38784.384109.2F. Epub 2006 Apr 7. PMID 16603564
- [Background] Eggli S, Kohlhof H, Zumstein M, Henle P, Hartel M, Evangelopoulos DS, Bonel H, Kohl S. Dynamic intraligamentary stabilization: novel technique for preserving the ruptured ACL. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1215-21. doi: 10.1007/s00167-014-2949-x. Epub 2014 Mar 21. PMID 24651979
- [Background] Gustavsson A, Neeter C, Thomee P, Silbernagel KG, Augustsson J, Thomee R, Karlsson J. A test battery for evaluating hop performance in patients with an ACL injury and patients who have undergone ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2006 Aug;14(8):778-88. doi: 10.1007/s00167-006-0045-6. Epub 2006 Mar 9. PMID 16525796
- [Background] Manske R, Reiman M. Functional performance testing for power and return to sports. Sports Health. 2013 May;5(3):244-50. doi: 10.1177/1941738113479925. PMID 24427396
- [Background] Itoh H, Kurosaka M, Yoshiya S, Ichihashi N, Mizuno K. Evaluation of functional deficits determined by four different hop tests in patients with anterior cruciate ligament deficiency. Knee Surg Sports Traumatol Arthrosc. 1998;6(4):241-5. doi: 10.1007/s001670050106. PMID 9826806
- [Background] Thomee R, Kaplan Y, Kvist J, Myklebust G, Risberg MA, Theisen D, Tsepis E, Werner S, Wondrasch B, Witvrouw E. Muscle strength and hop performance criteria prior to return to sports after ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2011 Nov;19(11):1798-805. doi: 10.1007/s00167-011-1669-8. Epub 2011 Sep 20. PMID 21932078
- [Background] Augustsson J, Thomee R, Karlsson J. Ability of a new hop test to determine functional deficits after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2004 Sep;12(5):350-6. doi: 10.1007/s00167-004-0518-4. Epub 2004 May 8. PMID 15138668
- [Background] Thomee R, Neeter C, Gustavsson A, Thomee P, Augustsson J, Eriksson B, Karlsson J. Variability in leg muscle power and hop performance after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2012 Jun;20(6):1143-51. doi: 10.1007/s00167-012-1912-y. Epub 2012 Feb 8. PMID 22314862
- [Background] Bjorklund K, Andersson L, Dalen N. Validity and responsiveness of the test of athletes with knee injuries: the new criterion based functional performance test instrument. Knee Surg Sports Traumatol Arthrosc. 2009 May;17(5):435-45. doi: 10.1007/s00167-008-0674-z. Epub 2008 Nov 28. PMID 19039577
- [Background] Reid A, Birmingham TB, Stratford PW, Alcock GK, Giffin JR. Hop testing provides a reliable and valid outcome measure during rehabilitation after anterior cruciate ligament reconstruction. Phys Ther. 2007 Mar;87(3):337-49. doi: 10.2522/ptj.20060143. Epub 2007 Feb 20. PMID 17311886
- [Background] Ageberg E, Thomee R, Neeter C, Silbernagel KG, Roos EM. Muscle strength and functional performance in patients with anterior cruciate ligament injury treated with training and surgical reconstruction or training only: a two to five-year followup. Arthritis Rheum. 2008 Dec 15;59(12):1773-9. doi: 10.1002/art.24066. PMID 19035430
- [Background] Abrams GD, Harris JD, Gupta AK, McCormick FM, Bush-Joseph CA, Verma NN, Cole BJ, Bach BR Jr. Functional Performance Testing After Anterior Cruciate Ligament Reconstruction: A Systematic Review. Orthop J Sports Med. 2014 Jan 21;2(1):2325967113518305. doi: 10.1177/2325967113518305. eCollection 2014 Jan. PMID 26535266
- [Background] Micheo W, Hernandez L, Seda C. Evaluation, management, rehabilitation, and prevention of anterior cruciate ligament injury: current concepts. PM R. 2010 Oct;2(10):935-44. doi: 10.1016/j.pmrj.2010.06.014. PMID 20970763